CLINICAL TRIAL: NCT04039698
Title: Monitoring of Hepatitis C Therapy Using Telemedicine in a Simplified Protocol With Pangenotypic Regimen in Non-cirrhotic Patients - a Single Group Clinical Trial in the National Public Health System in Brazil
Brief Title: Monitoring of Hepatitis C Treatment Using Telemedicine - a Clinical Trial in Public Health System in Brazil
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Ministry of Health, Brazil (Other Government); State Secretary of Health of Rio Grande do Sul (Unknown); TelessaúdeRS / UFRGS (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018-0290; Plataforma Brasil (CAAE) (Other: 91278418200005327)
Record Dates: First submitted 2019-07-30; First posted 2019-07-31 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C; Telemedicine; Direct acting antivirals; Public Health
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — Telemedicine; sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Telemedicine (Experimental): Sofosbuvir 400mg and velpatasvir 100mg qd for 12 weeks Telemedicine support
  Interventions: Other: Telemedicine; Drug: Velpatasvir/Sofosbuvir

INTERVENTIONS:
Other: Telemedicine — Telemedicine monitoring and teleconsultation by video calls
Drug: Velpatasvir/Sofosbuvir — Velpatasvir 100mg / Sofosbuvir 400mg once a day for twelve weeks
  Other Names: Epclusa

SUMMARY:
The study is a non-randomized, single group clinical trial on monitoring hepatitis C therapy using telemedicine. Patients with chronic hepatitis C without cirrhosis will be treated with the pangenotypic regimen of direct acting antivirals sofosbuvir and velpatasvir for 12 weeks after a single visit to the clinic, in which treatment will be prescribed. Patients will be then monitored by telemedicine tools, like instant message application, telephone and video calls and by his or her primary physician when needed. Twelve weeks after treatment conclusion, hepatitis C virus RNA levels will be measured on a blood sample, indicating the cure rate and efficacy of this protocol on HCV treatment.

The primary objective of the study is to address the feasibility and applicability of the usage of telemedicine tools to increase access and monitor HCV treatment with direct-acting antivirals in public health in Brazil.

DETAILED DESCRIPTION:
Scientific rationale

It's estimated that 0.7% of the Brazilian population is infected with hepatitis C virus (HCV). In March 2018, the Ministry of Health defined all patients with HCV to be able to receive direct-acting antivirals (DAAs) from the public health system without any charges. Though this "universal-access policy", frequently there are still many obstacles for patients to actually get at the treatment: patients living in cities distant from big centres and underserved by specialized physicians in the country, lack of medical doctors experienced in HCV treatment in the public system, delay between prescription and starting of medications because of administrative issues, and socioeconomic vulnerability among people.

Telemedicine tools are powerful ways of reaching people living distant from big centres, and there are some successful international experiences with hepatitis C treatment in this field, like Project ECHO® (Extension for Community Healthcare Outcomes). In Brazil, there is a national program, geographically located in Porto Alegre, that uses telemedicine to improve healthcare quality in primary care by offering continuous education and teleconsultations (by text or toll-free hotline) to community physicians and other healthcare professionals working in public primary care institutions all over the country.

Primary objective

To address the applicability of telemedicine tools to increase access and monitor HCV treatment with direct-acting antivirals in public health in Brazil.

Research methods

HCV-infected patients in the waiting list for specialized consultation with gastroenterologist or infectious disease physician will be recruited to a meeting that will consist of a HCV lecture followed by individual, focused consultation with medical history, analysis of previous lab results (including fibrosis evaluation by the AST-to-platelets ratio index - APRI) and collection of blood samples. All patients will receive a prescription of pan-genotypic DAA sofosbuvir and velpatasvir regimen for 12 weeks according to the Brazilian Ministry of Health's Treatment Protocol, along with orientations about use and potential side effects and ways to contact the telemedicine centre - mobile phone instant messages and WhatsApp® messages, phone calls and video calls. Issues regarding the administrative process will be held by the study team and medications will be delivered to each patient's city or region at the time they're available.

Before starting treatment, patients will be oriented about treatment administration, its potential side effects and ways of contacting the research team by text messages, phone calls and, when appropriate, teleconsultation by video teleconference with the patient and one of the healthcare professionals of the study. During the treatment course, adverse effects will be monitored and, when present, graded by the Division of AIDS (DAIDS) Table from the National Institutes of Health.

The family physicians working in each patient area will be oriented about this study and HCV treatment. Moreover, they will be invited to join the regular Project ECHO® meetings held by the Brazilian centre located at Porto Alegre. Healthcare professionals also have the toll-free hotline to get in touch with the telemedicine program and investigators. HCV-RNA will be collected 12 weeks after the end of therapy at a local institution next to patient home or city.

ELIGIBILITY:
Inclusion Criteria:

* Have voluntarily signed the informed consent form;
* Chronic hepatitis C confirmed by positive HCV-RNA;
* Have been referred to specialized consultation in gastroenterology or infectious disease in the Brazilian Public Health System in Porto Alegre;
* Have previous fibrosis staging (eg. liver biopsy, Fibroscan®) or laboratory tests for APRI score calculation.

Exclusion Criteria:

* Suspicion or diagnosis of cirrhosis based on:
* Hepatic elastography ≥12.5 kPa on Fibroscan®;
* APRI score ≥2.0;
* Clinical, ultrasound or endoscopic evidence of cirrhosis or portal hypertension;
* Previous HCV treatment with direct acting antivirals;
* HIV coinfection with antiretroviral treatment incompatible with HCV antivirals;
* Previous solid organ transplant;
* Significant comorbidity that may interfere with the HCV treatment
* Creatinine clearance < 30 mL/min;
* Platelets < 150.000/mL;
* Pregnant or breastfeeding female;
* Woman of childbearing age without use or that does not accept to use effective contraception during treatment and during the 30 days after treatment end;
* Inability or unwillingness to provide informed consent or abide by the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Sustained virologic response | 12 weeks post end of antiviral therapy (SVR12)
  Proportion of treated patients with undetectable hepatitis C virus RNA levels measured by a real time polymerase chain reaction (PCR) with a lower limit of detection ≤ 12 IU/mL

SECONDARY OUTCOMES:
Adherence to antiviral treatment | 12 weeks after antiviral treatment initiation
  Proportion of patients with treatment completion
Patient satisfaction with the treatment | 12 weeks post end of antiviral therapy (SVR12)
  Patient satisfaction with the telemedicine support measured by a a questionnaire applied to all participants
Adverse effects | 12 weeks post end of antiviral therapy (SVR12)
  Incidence of adverse effects related to treatment reported by patients
Severe adverse effects | 12 weeks post end of antiviral therapy (SVR12)
  Incidence of severe or life threatening (grade 3 or 4) adverse effects related to treatment reported by patients

OTHER OUTCOMES:
Rate of primary physicians participation after invitation to project ECHO® | 12 weeks post end of antiviral therapy (SVR12)
  To address the participation rate on Project ECHO® meetings of primary care physicians who referred patients enrolled in the study

CONTACTS AND LOCATIONS:
Overall Officials: Mario R Alvares-da-Silva, PhD, Study Chair — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
We plan to open data that might be useful for policy makers, specially in Brazil, and for researchers interested in replicate the study.
Supporting Information: Study Protocol, CSR
Time Frame: starting after the publication
Access Criteria: Researchers or public health policy makers interested in perform analyses to replicate the study or protocol of telemonitoring.

REFERENCES:
- [Derived] Oliveira JC, Schacher FC, Costa MB, Kolling MG, Costa RB, Scherer HC, Fernandes PM, Katz N, Goncalves MR, Rados DV, Alvares-da-Silva MR. TeleHCV: A single-visit protocol and minimal passive remote monitoring are sufficient to achieve high SVR with a sofosbuvir-velpatasvir regimen. Clinics (Sao Paulo). 2025 Apr 23;80:100643. doi: 10.1016/j.clinsp.2025.100643. eCollection 2025. PMID 40273497